CLINICAL TRIAL: NCT05719272
Title: HeadPulse Large Vessel Occlusion Validation Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: MindRhythm, Inc. (Industry)
Collaborators: University at Buffalo (Other); The Cooper Health System (Other)
Responsible Party: Sponsor
Other Study IDs: EPISODE_LVO_MR1
Record Dates: First submitted 2022-11-16; First posted 2023-02-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute ischemic stroke (AIS) is a treatable disease if patients can be transported and treated at stroke centers. MindRhythm, Inc (sponsor) has developed an investigational medical device that is designed for prehospital field use to differentiate the two major forms of acute ischemic stroke, namely Large Vessel Occlusion (LVO) stroke and non-large vessel occlusion stroke. The intended use is for paramedics to decide which destination hospital is best for the patient based on the device result. Large vessel occlusion stroke patients should be brought directly to comprehensive stroke centers which can perform thrombectomy, and non-large vessel occlusion stroke should be brought to primary stroke centers. Use of the device will save time getting the patient to thrombectomy and all others to intravenous thrombolytics or blood thinners that clear clots improves outcomes for all patients.

The Harmony 5000 device manufactured by MindRhythm has been tested in the pre-hospital environment, but because large vessel occlusion stroke is less common than non-large vessel occlusion stroke, the sponsor wants to obtain additional recordings from patients with large vessel occlusion to better refine their algorithms. Investigators will perform acute recordings on patients who arrive at the medical center who have computed tomography angiography studies showing the presence of large vessel occlusion stroke stroke, and on patients transferred to the angiography suite for thrombectomy. Recordings are performed in parallel to standard workflow of large vessel occlusion stroke patients so the research will not delay treatments.

DETAILED DESCRIPTION:
Eligible participants will be 18 years of age plus with known large vessel occlusion who have been transferred to the emergency department. Recordings can be made just prior to the thrombectomy or within 2 hours of computed tomography angiography and no thrombectomy performed.

Participants will be excluded if they have an open wound on the scalp or are prisoners.

The MindRhythm Harmony headset will be placed on the subject (a total of 50 subjects) along with ECG leads and a 3 minute recording of the HeadPulse (cranial waveform) will be performed while the subject remains as still as possible. The data will then be transferred to MindRhythm for analysis and ultimate improvement of the diagnostic stroke algorithm.

ELIGIBILITY:
Inclusion Criteria:

* adult patient Known LVO (transferred or arrived at our ED) ICA-T, M1, M2 or Basilar Artery Recording can be made just prior to thrombectomy, or within 2 hours of CTA and no thrombectomy performed

Exclusion Criteria:

* Prisoner Open scalp wound

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill patients who have experienced and have a confirmed ischemic stroke of the most critical type: a large vessel occlusion who are admitted to the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-16 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
HeadPulse Waveform Data | 90 seconds
  Waveform data associated with the changes in brain function as a result of the cranial effect of the. cardiac cycle

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lovoi, PhD, Principal Investigator — CTO of Sponsor
Locations (2):
- United States (2):
  - Cooper University Hospital, Camden, New Jersey
  - University at Buffalo, Buffalo, New York

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT05719272/Prot_000.pdf
  • Informed Consent Form (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT05719272/ICF_001.pdf